CLINICAL TRIAL: NCT07072416
Title: Aquatic Based Exercises Versus Mirror Therapy on Hand Dexterity and Strength in Hemiplegic Child
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Alaa Noureldeen Kora (Other)
Responsible Party: Sponsor-Investigator, Alaa Noureldeen Kora, Assistant Professor, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P.T.REC/012/005354
Record Dates: First submitted 2025-07-09; First posted 2025-07-18 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Cerebral Palsy (CP); Hemiplegia and Hemiparesis
Keywords: Aquatic Based Exercises; Hemiplegic Child; Hand Dexterity; Mirror Therapy; Hand Strenght; Cerebral Palsy
MeSH Terms: conditions — Cerebral Palsy; Hemiplegia; Paresis | interventions — Aquatic Therapy; Mirror Movement Therapy

STUDY DESIGN:
Intervention Model Description: Randomized Controlled Trial
Who Masked: Outcomes Assessor
Masking Description: Blinding to the assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1: Aquatic Therapy (Experimental): Children in Group A will receive aquatic based exercises and a designed physical therapy program
  Interventions: Other: Aquatic Exercise; Other: Designed physical therapy program.
- Group 2: Mirror Therapy (Experimental): Group B will receive mirror therapy and a designed physical therapy program
  Interventions: Other: Mirror Therapy; Other: Designed physical therapy program.
- Group 3: Control Group (Other): Control Group (C) will receive a designed physical therapy program.
  Interventions: Other: Designed physical therapy program.

INTERVENTIONS:
Other: Aquatic Exercise — Aquatic exercise or hydrotherapy, involving the performance of physical exercise in water, has been determined to have an assortment of beneficial health impacts on healthy individuals and those with chronic diseases. Aquatic exercise has been determined to enhance strength, balance, flexibility, and the quality of life, particularly among groups like postmenopausal women, patients with osteoarthritis, Parkinson's disease, and type 2 diabetes
  Arms: Group 1: Aquatic Therapy
Other: Mirror Therapy — Mirror therapy is a type of rehabilitation where visual feedback is employed to induce movement and recovery in an affected limb by asking the patients to observe the reflection of their healthy limb in a mirror, giving the illusion that both limbs are moving normally.
  Arms: Group 2: Mirror Therapy
Other: Designed physical therapy program. — The program will start with 10 minutes of poolside exercises including warming up, active range of motion and stretching followed by 20 minutes of aquatic exercise in the pool. The pool session consists of 20 minutes of active range of motion, stretching and strengthening exercises

SUMMARY:
Cerebral palsy (CP) is a neurologic disorder that affects motor function, balance, and posture, and spastic hemiplegia is found in about one-third of persons with CP and often leads to devastating upper limb disability. Rehabilitation interventions such as aquatic therapy and mirror therapy are commonly utilized to improve motor function and functional independence. Water therapy takes advantage of water resistance and buoyancy to relax tightened muscles, promote gross motor function, and increase muscle endurance and strength with studies showing significant improvements in motor skills as well as a reduction in spasticity in CP children, especially hemiplegic children. Water therapy can also be more enjoyable and convenient for kids, but safety has to be considered. Mirror therapy does utilize visual feedback, but to cause the movement in the paralyzed limb, and can increase hand dexterity and grip strength by stimulating the neural pathways through the illusion of movement. Although aquatic therapy has shown well-defined advantages in motor functioning and muscle tone, comparison of the efficacy of aquatic exercises and mirror therapy for hand dexterity and grip strength in hemiplegic CP has been limited, and further studies are indicated to establish their relative merits and potential complementary uses.

DETAILED DESCRIPTION:
Cerebral palsy (CP) is a neurological impairment of motor disorder, balance, movement disorder, and postural deformities that appear during infancy and early childhood, although muscle tone and posture related abnormalities becomes more prominent in later years . Globally CP occurs 1.5 to more than 4 per 1000 live births.

One of the types of CP is spastic hemiplegia, known as half-body paralysis and the prevalence is about 35.1% of all children with CP . Upper limb function impairment is a common and disability consequence of problems in reaching, pointing, and taking, releasing and manipulating objects . The ability to reach and grasp things is one of the basic tasks in activities of daily living.

Multiple approaches in the physical therapy are being used in the rehabilitation of CP such as stretching, strengthening, Neuro-developmental technique (NDT), motor relearning programs in reducing the spasticity and improving functional level in CP (Dimitrijević et al., 2012). During current practices, primary focus on improving the functional independency and motor skills, thus aquatic therapy is good approach in this regard (Declerck et al., 2013).

Furthermore, hydrotherapy is effective treatment mode due to buoyancy and hydrostatic properties of water. Buoyancy force is equal to the weight of the fluid displaced by the object. According the hydrotherapy is an effective treatment option in CP due to its thermal and mechanical effects.

Thermal effects relax the muscle and facilitates in reducing the spasticity while mechanical effects of water are sufficient in reducing the effect of gravity and minimizing the joint loading, furthermore, water provides enjoyable environment to perform multiple functional activities for cerebral palsy (Getz et al., 2012). Exercises in the pool are always performed at the temperature of 33°- 35oC that is essential in reducing the spasticity by relaxing the muscles (Adar et al., 2017). Besides these effects hydrotherapy has effects on strengthening the muscles and endurance since water creates resistance during walking that strengthens the muscles (Khalaji et al., 2017). Activities performed in water are easier and effective as compared to the land but it has a major safety issue that should be identified before the start of exercises for the better results (Adar et al., 2017). Hydrotherapy has several positive effects in the management of spasticity, joint range of motion and improving balance in CP. Since the aquatic exercise reduces spasticity thus has potential effects in improving the gross motor functions among CP.

Among non-invasive approaches, mirror therapy is a relatively new approach that focuses on visual stimulation and the movements of limbs without damage. The reflection of the healthy limb movement in the mirror is thought the affected limb is moving naturally (Fukumura et al., 2007). In this method, the patient places his hands on the two sides of the mirror. Thus, the patient understands the reflection of his healthy hand in the mirror as his affected hand (Mc Cabe et al., 2008).

Statement of problem:

Is there difference between effects of aquatic based exercises and mirror therapy on hand dexterity and hand grip strength in children with hemiplegic cerebral palsy?

Purpose of study:

The purpose of this study is:

* To investigate the effect of aquatic based exercises and mirror therapy on hand dexterity and hand grip strength in children with hemiplegic cerebral palsy
* To investigate the correlations between the effects of aquatic based exercises, mirror therapy and control group on hand dexterity and hand grip strength in children with hemiplegic cerebral palsy.

ELIGIBILITY:
Inclusion Criteria:

* Children with Hemiplegic cerebral palsy
* Children with mild to moderate spasticity of wrist muscles spasticity will range between (0-4) score according to Modified Ashworth Scale.
* Children will be able to follow the instructions.
* Children without any genetic disorders.

Exclusion Criteria:

* Cognitive impairment.
* Unilateral neglect disorders.
* Orthopedic dysfunction.
* Visual impairment.
* Verbal impairment.
* Open wound or infection
* Fixed contractures.
* Previous limb surgeries within 6 months.
* Resting angina.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 45 (Actual)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-08-30 (Estimated); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
Box and Block Test: It was used to assess gross manual dexterity | 3 Months
  The Box and Block Test (BBT) is a widely used test to evaluate gross manual dexterity by rehabilitation centers and occupational therapy clinics. The individual has to move as many blocks as possible from one of the compartments of a box to the other in a given time period, usually one minute, using one hand at a time. The BBT is valued for simplicity, ease of use, and strong reliability and validity across the lifespan, and in clinical populations like children, adults, and those with neurological or musculoskeletal disorder
Hand held dynamometer to assess hand grip strength. | 3 Months
  A popular, trustworthy, and legitimate tool for evaluating hand grip strength-a crucial sign of general muscle function and health-is a hand-held dynamometer.

CONTACTS AND LOCATIONS:
Locations (1):
- Damanhur Medical National Institute Hospital, Damanhur, Beheira, Egypt

IPD SHARING:
Plan to Share IPD: No
It will provided only upon reasonable request

REFERENCES:
- [Background] Adar S, Dundar U, Demirdal US, Ulasli AM, Toktas H, Solak O. The effect of aquatic exercise on spasticity, quality of life, and motor function in cerebral palsy. Turk J Phys Med Rehabil. 2017 Aug 14;63(3):239-248. doi: 10.5606/tftrd.2017.280. eCollection 2017 Jun. PMID 31453460
- [Background] Roostaei M, Baharlouei H, Azadi H, Fragala-Pinkham MA. Effects of Aquatic Intervention on Gross Motor Skills in Children with Cerebral Palsy: A Systematic Review. Phys Occup Ther Pediatr. 2017 Oct 20;37(5):496-515. doi: 10.1080/01942638.2016.1247938. Epub 2016 Dec 14. PMID 27967298
- [Background] El-Shamy SM. Effects of Antigravity Treadmill Training on Gait, Balance, and Fall Risk in Children With Diplegic Cerebral Palsy. Am J Phys Med Rehabil. 2017 Nov;96(11):809-815. doi: 10.1097/PHM.0000000000000752. PMID 28410250
- [Background] Lai CJ, Liu WY, Yang TF, Chen CL, Wu CY, Chan RC. Pediatric aquatic therapy on motor function and enjoyment in children diagnosed with cerebral palsy of various motor severities. J Child Neurol. 2015 Feb;30(2):200-8. doi: 10.1177/0883073814535491. Epub 2014 Jun 5. PMID 24907137
- [Background] Ryu K, Ali A, Kwon M, Lee C, Kim Y, Lee G, Kim J. Effects of assisted aquatic movement and horseback riding therapies on emotion and brain activation in patients with cerebral palsy. J Phys Ther Sci. 2016 Dec;28(12):3283-3287. doi: 10.1589/jpts.28.3283. Epub 2016 Dec 27. PMID 28174435
- [Background] Stavsky M, Mor O, Mastrolia SA, Greenbaum S, Than NG, Erez O. Cerebral Palsy-Trends in Epidemiology and Recent Development in Prenatal Mechanisms of Disease, Treatment, and Prevention. Front Pediatr. 2017 Feb 13;5:21. doi: 10.3389/fped.2017.00021. eCollection 2017. PMID 28243583